CLINICAL TRIAL: NCT00411346
Title: Nurse-Led Telemonitoring Programme in Asthmatic Outpatients: a Randomized Controlled Trial
Brief Title: Patient Research In Self-Management of Asthma (PRISMA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 02-157.1
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2006-12-14 (Estimated); Status verified 2006-12

CONDITIONS: Asthma
Keywords: Asthma; Self-Monitoring; Cost-effectiveness
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Procedure: Nurse-led telemonitoring

SUMMARY:
The objective of this study was to investigate if a nurse-led telemonitoring programme is effective and cost-effective in asthmatic outpatients, aged seven years and older.

DETAILED DESCRIPTION:
At the present day asthma is one of the most common chronic illnesses worldwide and the prevalence is still increasing. Asthma can be treated and controlled with guidance of health care professionals, and self-monitoring is an important aspect in this control.

Respiratory nurses have become common caregivers in the treatment and control of asthma. Advances in information and communication technology have created the potential to monitor the asthma status of patients at a distance, named telemonitoring. These two developments come together in nurse-led telemonitoring programmes. Lung function tests, from which the peak expiratory flow (PEF) is the most commonly used, are recorded into an electronic monitor. By transferring monitor data to a central database a nurse can continuously supervise the disease status of individual patients. The use of stepwise protocols can enable nurses to independently adjust the medication by one step.

Design: Randomized controlled trial comparing a nurse-led telemonitoring programme versus regular care in asthmatic outpatients aged 7 years and older.

Primary outcome parameter: asthma-specific quality of life. Secondary outcome parameters: symptoms, generic quality of life, direct and indirect costs, satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 7 years or older
* Asthma severity of stage I - III as described in the GINA guidelines
* Must be competent to use an asthma monitor
* Must possess a household phone connection

Exclusion Criteria:

* Respiratory co-morbidity

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112
Dates: Start 2003-01; Study Completion 2004-11

PRIMARY OUTCOMES:
Asthma-specific quality of life at one year.

SECONDARY OUTCOMES:
Asthma symptoms at one year
generic quality of life at one year
direct and indirect costs during one year
satisfaction with and feasibility of the intervention at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Emiel FM Wouters, MD PhD, Study Chair — Department of Respiratory Medicine
Locations (1):
- University Hospital Maastricht, Maastricht, Limburg, Netherlands